CLINICAL TRIAL: NCT01547091
Title: Clinical Trial of Umbilical Cord-Derived Mesenchymal Stem Cells Transplantation for Rheumatoid Arthritis-Phase I/II
Brief Title: Safety and Efficacy Study of Umbilical Cord-Derived Mesenchymal Stem Cells for Rheumatoid Arthritis
Acronym: RA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alliancells Bioscience Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alliancells-1
Record Dates: First submitted 2012-02-22; First posted 2012-03-07 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Mesenchymal Stem Cells; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- UC-MSCs Treatment (Experimental): Patients in UC-MSCs treatment will be infused umbilical cord-derived mesenchymal stem cells intravenously only.
  Interventions: Biological: Umbilical Cord-Derived Mesenchymal Stem Cells (UC-MSCs)
- DMARDS (Active Comparator): Patients will be treated by Rheumatoid Arthritis With Disease-Modifying Drugs (DMARDs).
  Interventions: Drug: Rheumatoid Arthritis With Disease-Modifying Drugs (DMARDs)
- UC-MSC+DMARDS (Active Comparator): Patients will be treated in combination with UC-MSC and DMARDS.
  Interventions: Biological: UC-MSC+DMARDS

INTERVENTIONS:
Biological: Umbilical Cord-Derived Mesenchymal Stem Cells (UC-MSCs) — -The UC-MSCs will be infused intravenously(single dose, 4x10^7 cells).The interval time is 3 months, and the study lasts for 12 months with 4 times infusion.
  Arms: UC-MSCs Treatment
Drug: Rheumatoid Arthritis With Disease-Modifying Drugs (DMARDs) — -Patients will be treated by conventional drugs (DMARDS) for alleviating disease.
  Arms: DMARDS
Biological: UC-MSC+DMARDS — The UC-MSCs will be infused intravenously(single dose, 4x10^7 cells).The interval time is 3 months, and the study lasts for 12 months with 4 times infusion.Meanwhile,patients will be treated by conventionally drugs if the disease is still not alleviated.
  Arms: UC-MSC+DMARDS

SUMMARY:
Rheumatoid arthritis is a chronic systemic disease, which is characterized by chronic inflammation in the synovial tissue. Rheumatoid arthritis will eventually result in the destruction of cartilage, bone and ligaments and joint deformity. The underlying hypothesis is that umbilical cord-derived mesenchymal stem cell (UC-MSCs) has anti-inflammatory effects and thus potentially alleviates the progression of rheumatoid arthritis. The study is to explore the safety and efficacy of UC-MSCs transplantation in treatment of rheumatoid arthritis.

DETAILED DESCRIPTION:
This study was supported by the National Natural Science Foundation of China (30872618)，The Shanxi Province Social Development Public Relations Project (2012K13-02-35), and The Military Medicine and Public Health Plan (CLZ120GA23)

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the classification criteria (2010) for rheumatoid arthritis, man or woman aged from 18 to 70 years old.
* Patients must be informed of the investigational nature of this study and give written informed consent in accordance with the institutional and hospital guidelines.
* Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on this trial. Women of child-bearing potential must have a pregnancy test performed within 72 hours prior to initiation of treatment.

Exclusion Criteria:

* Any history of ongoing, significant or recurring infections.
* Any active inflammatory diseases other than RA.
* Significant cardiac or pulmonary disease.
* End-stage renal failure.
* Pregnant or nursing women may not participate due to the possibility of fetal harm or harm to nursing infants from this treatment regimen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Safety of MSC treatment. | six months
  Adverse Events will be recorded in a patient or clinical investigation subject who administers MSC and will be evaluated a causal relationship with the treatment.

SECONDARY OUTCOMES:
RA Serology | 1, 3 and 6 months
  Rheumatoid Factor, C-reactive protein
Disease Activity Score (DAS 28) Index Mean Change From Baseline | 1, 3 and 6 months
Patient's assessment of pain. | 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mingyuan Wu, MD,PhD, Principal Investigator — Eastern Union Stem Cell & Gene Engineering Co.,Ltd，Alliancells Biosciences Co., Ltd; Yongjun Liu, MD,PhD, Principal Investigator — Alliancells Biosciences Co., Ltd; Liming Wang, MD, Study Director — The 323 Hospital of Chinese People's Liberation Army; Haijie Ji, MD, Principal Investigator — Alliancells Biosciences Co., Ltd.
Locations (1):
- The 323 Hospital of Chinese People's Liberation Army, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Wang H, Wu M, Liu Y. Are mesenchymal stem cells major sources of safe signals in immune system? Cell Immunol. 2012;272(2):112-6. doi: 10.1016/j.cellimm.2011.10.010. Epub 2011 Oct 29. PMID 22138499
- [Background] Wang L, Ji H, Zhou J, Xie J, Zhong Z, Li M, Bai W, Li N, Zhang Z, Wang X, Zhu D, Liu Y, Wu M. Therapeutic potential of umbilical cord mesenchymal stromal cells transplantation for cerebral palsy: a case report. Case Rep Transplant. 2013;2013:146347. doi: 10.1155/2013/146347. Epub 2013 Mar 3. PMID 23533920